CLINICAL TRIAL: NCT04661618
Title: A Randomized-Control Study of Gym Tonic's Community Based Strength Training Intervention on Physical Function and Frailty Reversal, for Elderly Singaporeans.
Brief Title: A Randomized-Control Study of Gym Tonic's Community Based Strength Training Intervention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseSync Pte Ltd (Industry)
Collaborators: Singapore Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GT/RCT/2018/001
Record Dates: First submitted 2020-11-19; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Frailty; Muscle Loss; Sarcopenia
MeSH Terms: conditions — Frailty; Muscular Atrophy; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomised-Control Trial
Who Masked: Investigator
Masking Description: Data is anonymized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GT (Active Comparator): 12 weeks of progressive training in the first phase and 12 weeks of maintenance training in the second phase.
  Interventions: Device: Gym Tonic programme and Gym equipment
- Control (Other): No intervention for the first phase and will be active comparator in the second phase.
  No intervention for the first 12 weeks (first phase) and 12 weeks of progressive training in the second phase.
  Interventions: Device: Gym Tonic programme and Gym equipment

INTERVENTIONS:
Device: Gym Tonic programme and Gym equipment — 12 week progressive training - Strength exercises on 6 pneumatic gym equipment following Gym Tonic's protocol twice a week 12 weeks maintenance training - Strength exercises on 6 pneumatic gym equipment following Gym Tonic's protocol once a week

SUMMARY:
Launched in April 2015 , Gym Tonic is the first of its kind cross-border exercise-as-medicine partnership between research institutions, business enterprises and service providers from Singapore and Finland. What sets Gym Tonic apart from other exercise programmes is its singular focus on strength training, necessary for frailty prevention and maintenance of functional independence for the elderly.

This randomized-control trial is to validate the Gym Tonic programme and data as well measuring its effectiveness in improving physical functions and reversing frailty.

DETAILED DESCRIPTION:
The RCT is conducted in 3 eldercare community centers. In each center, a group of elderly will be randomly sorted into 2 groups. An intervention group and a control group.

The intervention group will go through 12 weeks of Gym Tonic progressive training programme. While the control group acts as a control. After the first 12 weeks, the intervention group will be going through another 12 weeks of Gym Tonic maintenance programme, while the control group will be going through the Gym Tonic progressive training programme.

Measurements of physical functions, isometric strength and frailty will be conducted pre trial, post 12 weeks and post 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and above
* Pre-frail or mildly frail, as measured by the 5 CHS criteria of physical frailty: unintentional weight loss, slowness, weakness, exhaustion, low activity level or FRAIL
* Able to ambulate without personal assistance
* Enrolled into the 3 sites above

Exclusion Criteria:

* Bedbound
* Terminally ill patients with life expectancy <12 months
* Significant cognitive impairment
* Major depression
* Wear pacemaker
* Severe audiovisual impairment
* Any progressive, degenerative neurologic disease
* Participating in other interventional studies
* Unavailable to participate for the full duration of the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 318 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Isometric Muscle Strength (Knee Extension) | week 0, week 12, week 24
  Measured via isometric performance recorder fixed to exercise machine for the right and left leg.
Change in Isometric Muscle Strength (Knee Flexion) | week 0, week 12, week 24
  Measured via isometric performance recorder fixed to exercise machine for the right and left leg.
Change in Isometric Muscle Strength (Hip Abduction) | week 0, week 12, week 24
  Measured via isometric performance recorder fixed to exercise machine for the above mentioned movement.
Change in Isometric Muscle Strength (Hip Adduction) | week 0, week 12, week 24
  Measured via isometric performance recorder fixed to exercise machine for the above mentioned movement.
Handgrip Strength | week 0, week 12, week 24
  Subject will be seated, with the arm unsupported, elbow joint at 90 degrees and wrist in a neutral position while holding the hand dynamometer.
  Subject would be required to squeeze the grip with maximum strength upon command for three attempts. The best result would be recorded.
SPPB Balance Test - Feet together (side-by-side) | week 0, week 12, week 24
  To balance in the said position for 10 seconds.
  Scored point will be determined by number of seconds held.
SPPB Balance Test - Semi-Tandem stand | week 0, week 12, week 24
  To balance in the said position for 10 seconds.
  Scored point will be determined by number of seconds held.
SPPB Balance Test - Tandem stand | week 0, week 12, week 24
  To balance in the said position for 10 seconds.
  Scored point will be determined by number of seconds held.
SPPB 5 times sit-to-stand | week 0, week 12, week 24
  Seated with arms folded across chest and with their back against the chair, Stand up fully and sit down fully with the back against the chair as quickly as possible.
  Scored point will be determined by the time to completely finish 5 repetitions.
SPPB Speed Walk Test (Normal) | week 0, week 12, week 24
  To walk 4 metres at participant's usual speed, scored point will be determined based on time taken to complete the 4-Metre walk.
SPPB Speed Walk Test (Fast) | week 0, week 12, week 24
  To walk 4 metres at participant's fastest speed, scored point will be determined based on time taken to complete the 4-Metre walk.

CONTACTS AND LOCATIONS:
Locations (1):
- PulseSync, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Goh A, Tan K, Choo PL, Ong PH, Wong WP, Wee SL. Effectiveness of a community-delivered pneumatic machine resistance training programme (Gym Tonic) for older adults at neighbourhood senior centres - a randomized controlled trial. Eur Rev Aging Phys Act. 2021 Oct 7;18(1):21. doi: 10.1186/s11556-021-00273-x. PMID 34620081
- See also: Promotional website for the Gym Tonic Programme. — http://www.gymtonic.sg